CLINICAL TRIAL: NCT05306717
Title: Impact of the Preventive Emotions Management Questionnaire on the Rates of Isolation and Mechanical Restraint Measures in the Psychiatric Admission Unit
Acronym: PACT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Charles Perrens, Bordeaux (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-A03039-32
Record Dates: First submitted 2022-03-14; First posted 2022-04-01 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Psychiatric Disorder
Keywords: Psychiatric Disorder; Prevention; Mechanical restraint; Isolation
MeSH Terms: conditions — Mental Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Epidemiology: The study will compare the rates of isolation and restraint of the two sectoral admission units welcoming people in care without consent for a period of one year.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — The study will compare the rates of isolation and restraint of the two sectoral admission units welcoming people in care without consent for a period of one year. The impact of the QPGE on the satisfaction scores will be systematically evaluated by a self-questionnaire for patients at the end of hospitalization. The QPGE is administered by a nurse during the reception interview of the patient in the unit.

SUMMARY:
This observational study assesses whether the use of the QPGE has an impact on the rates of isolation and mechanical restraint in adult psychiatric admission units. It is supplemented by a qualitative survey that will collect the experience of caregivers using the QPGE.

DETAILED DESCRIPTION:
The use of isolation and mechanical restraint in psychiatry has deleterious consequences for the patient. Caregivers also testify to their dissatisfaction with using these methods. The Coping Agreement Questionnaire (CAQ) is a form presented to the patient admitted to a psychiatric unit in the United States that has shown a significant effect on the reduction of coercive measures. It has been translated into French under the name Questionnaire Préventif de la Gestion des Emotions (QPGE). In France, the Haute Autorité de Santé has been recommending this type of tool since 2016 in the form of shared prevention plans to better prevent moments of violence.

The main objective is to assess whether the use of a shared prevention plan based on the Preventive Emotions Management Questionnaire (QPGE) can reduce the rates of isolation measures and mechanical restraint in hospitalized people. in a sectoral admission unit receiving patients in care without consent.

ELIGIBILITY:
Inclusion Criteria:

* Have been hospitalized in psychiatric admission unit with an entry date between January 1, 2020 and December 31, 2020
* Be at least 18 years old at the time of hospitalization
* Master the French language in order to have benefited from the QPGE and the satisfaction questionnaire

Exclusion Criteria:

* Being the subject of an isolation and/or restraint measure, decided in another unit before, during the transfer to the study places
* To have objected to the use of data collected during hospitalization following the information in the welcome booklet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with psychiatric disorders and hospitalized in a sectoral admission unit receiving patients in care without consent
Sampling Method: Non-Probability Sample
Enrollment: 416 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of isolation measures.(%) | up to 1 year
  Isolation and/or restraint notified in the registers dedicated to the monitoring of measures restricting liberty in the admission units during the study period
Rate of restraint measures.(%) | up to 1 year
  Isolation and/or restraint notified in the registers dedicated to the monitoring of measures restricting liberty in the admission units during the study period

SECONDARY OUTCOMES:
Rate of isolation measures not associated with an episode of mechanical restraint (%) | up to 1 year
Duration of isolation measures not associated with an episode of mechanical restraint. (hours) | up to 1 year
Rate of mechanical restraint measures (%) | up to 1 year
Duration of mechanical restraint measures (hours) | up to 1 year
User satisfaction score at the end of hospitalization | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Vincent BILLE, Study Director — Advanced Practice Nurse
Locations (1):
- Centre Hospitalier Charles Perrens, Bordeaux, Gironde, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Beghi M, Peroni F, Gabola P, Rossetti A, Cornaggia CM. Prevalence and risk factors for the use of restraint in psychiatry: a systematic review. Riv Psichiatr. 2013 Jan-Feb;48(1):10-22. doi: 10.1708/1228.13611. PMID 23438697
- [Result] Riahi S, Thomson G, Duxbury J. An integrative review exploring decision-making factors influencing mental health nurses in the use of restraint. J Psychiatr Ment Health Nurs. 2016 Mar;23(2):116-28. doi: 10.1111/jpm.12285. Epub 2016 Jan 26. PMID 26809740
- [Result] Bowers L, Allan T, Simpson A, Nijman H, Warren J. Adverse incidents, patient flow and nursing workforce variables on acute psychiatric wards: the Tompkins Acute Ward Study. Int J Soc Psychiatry. 2007 Jan;53(1):75-84. doi: 10.1177/0020764007075011. PMID 17333953
- [Result] Bowers L, Alexander J, Bilgin H, Botha M, Dack C, James K, Jarrett M, Jeffery D, Nijman H, Owiti JA, Papadopoulos C, Ross J, Wright S, Stewart D. Safewards: the empirical basis of the model and a critical appraisal. J Psychiatr Ment Health Nurs. 2014 May;21(4):354-64. doi: 10.1111/jpm.12085. Epub 2014 Jan 24. PMID 24460906